CLINICAL TRIAL: NCT02765633
Title: A Prospective, Open-Label, Single-Arm, Multi-Center Study To Assess The Pharmacokinetics/Pharmacodynamics (PK/PD) And Safety Of Different Cangrelor Doses In Neonatal Subjects At Risk Of Thrombosis
Brief Title: Cangrelor Neonatal PK/PD and Safety Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MDCO-CAN-15-01; 2016-000134-22 (EudraCT Number)
Record Dates: First submitted 2016-04-14; First posted 2016-05-06 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Partial Obstruction of Systemic to Pulmonary Artery Shunt; Complete Obstruction of Systemic to Pulmonary Artery Shunt
MeSH Terms: interventions — cangrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cangrelor (Experimental): Cangrelor in up to four (4) dose cohorts consisting of a minimum of five participants in each cohort. One cohort of five participants will be enrolled at a time. Cohort 1 subjects will receive Cangrelor at 0.5 mcg/kg/min. Cohort 2 subjects will receive Cangrelor at 0.25 mcg/kg/min. Subsequent cohort dosing decisions are made at the completion of enrollment in each cohort.
  Interventions: Drug: Cangrelor

INTERVENTIONS:
Drug: Cangrelor

SUMMARY:
The purpose of this study is to assess the PK/PD and safety profile of cangrelor in neonatal participants at risk of thrombosis.

ELIGIBILITY:
Inclusion criteria:

1. Males and females with congenital heart disease, and ranging in age from birth through 28 days of life
2. Postoperative neonatal cardiac participants with placement of systemic-to-pulmonary artery palliative shunts, right ventricle to pulmonary artery palliative shunts, or ductus arteriosus stents who are at risk of thrombotic events after repair for structural congenital heart disease.
3. Written informed consent from a parent/legal guardian
4. Life expectancy of at least 15 days at study entry

Participants will be excluded from the study if any of the following exclusion criteria apply:

1. History of intracerebral bleed (confirmed by a ultrasound (US) of the head prior to surgery), or cerebral arteriovenous malformation, or any prior bleed with neurological deficit
2. Gastrointestinal or urinary bleeding
3. Cerebrovascular accident or any cerebrovascular accident with a residual neurological deficit
4. Known congenital or acquired bleeding or clotting disorder
5. Weight less than 2.5 kilograms (kg)
6. Adjusted gestational age less than 37 weeks
7. Platelet count less than 100,000 cells/microliter (µL)
8. Chest and/or mediastinal tube blood output of greater than 3 milliliters (mL)/kg/hour (hr) at the time of cangrelor administration
9. Participants with evidence of severe hepatic or renal failure [aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than three times normal for age or total bilirubin greater than 20 milligrams (mg)/deciliter (dL); creatinine greater than 2 times the normal upper limit]
10. Known allergy to cangrelor or known sensitivity to any component of cangrelor
11. Any condition that in the investigator's opinion would constitute a contraindication to participation in the study or cause inability to comply with the study requirements
12. Participation in another investigational therapeutic drug or investigational therapeutic device trial within 30 days of starting study
13. Participants who have been receiving warfarin (Coumadin®) therapy

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Total plasma concentrations of cangrelor and its primary metabolite, AR C69712, during administration and after cessation of the infusion in neonates | During study drug infusion through 8 hours post infusion
Proportion of participants in each cohort who achieve ≥90% inhibition of final platelet aggregation as measured by light transmittance aggregometry (LTA) using 20 micromolar (µM) adenosine diphosphate (ADP) in platelet rich plasma | During study drug infusion through 1 hour post infusion
Individual recovery of platelet function in neonates after cessation of the infusion | Up to 1 hour post infusion
Assessment of the safety of cangrelor in neonatal participants by evaluating adverse events (AEs) and serious adverse events (SAEs) | from start of cangrelor infusion through 48 hours post cangrelor infusion

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Diacovo, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Medical Center, New York, New York
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vargas D, Zhou H, Yu X, Diamond S, Yeh J, Allada V, Krishnamurthy G, Price M, Allen B, Alexander J, Schmidhofer J, Kreutzer J, Vincent J, Morell V, Bacha E, Diacovo T. Cangrelor PK/PD analysis in post-operative neonatal cardiac patients at risk for thrombosis. J Thromb Haemost. 2021 Jan;19(1):202-211. doi: 10.1111/jth.15141. Epub 2020 Nov 29. PMID 33078501
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2016-000134-22/results